CLINICAL TRIAL: NCT01783847
Title: Study of Visual Recovery After Erythropoietin (EPO) Injection, in Patients With Traumatic Optic Neuropathy (TON)
Brief Title: Traumatic Optic Neuropathy Treatment Trial (TONTT)
Acronym: TONTT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Iran University of Medical Sciences (Other); Mashhad University of Medical Sciences (Other); Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 90-01-124-12972
Record Dates: First submitted 2013-02-01; First posted 2013-02-05 (Estimated); Results first posted 2018-09-12 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2016-04

CONDITIONS: Traumatic Optic Neuropathy
Keywords: Erythropoietin; Traumatic Optic Neuropathy; Visual function
MeSH Terms: conditions — Optic Nerve Injuries | interventions — Observation; Methylprednisolone Acetate

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Recombinant human erythropoietin (EPO) (Experimental): Intravenous EPO 10,000 IU for 5-13 years of age and 20,000 IU for >13 years/ day for 3 days
  Interventions: Drug: Recombinant human erythropoietin (EPO)
- Methylprednisolone (Active Comparator): Just Intravenous Methyl prednisolone 250 mg every 6 hours for 3 days.
  Interventions: Drug: Methyl prednisolone
- Observation (Other): Observation
  Interventions: Other: Observation

INTERVENTIONS:
Drug: Recombinant human erythropoietin (EPO) — 4000 units per vial
  Other Names: EPO (Pooyesh darou Co., Tehran)
  Arms: Recombinant human erythropoietin (EPO)
Other: Observation — Just observation
  Arms: Observation
Drug: Methyl prednisolone — 250 mg every 6 hours for 3 days.
  Other Names: Depo-Medrol
  Arms: Methylprednisolone

SUMMARY:
The pathophysiology of Traumatic Optic Neuropathy (TON) is thought to be multifactorial, and some researchers have also postulated a primary and secondary mechanism of injury.TON is categorized as direct or indirect.In indirect TON cases, the injury to the axons is thought to be induced by shearing forces that are transmitted to the fibers or to the vascular supply of the nerve. Studies have shown that forces applied to the frontal bone and malar eminences are transferred and concentrated in the area near the optic canal. The tight adherence of the optic nerve's dural sheath to the periosteum within the optic canal is also thought to contribute to this segment of the nerve being extremely susceptible to the deformative stresses of the skull bones. Such injury leads to ischemic injury to the axons of the retinal ganglion cells within the optic canal. At present, no studies validate a particular approach to the management of TON. There are three management lines for these patients that include 1)observation only;2)medical treatment with high or megadoses of methylprednisolone; and 3)surgical intervention. Generally no line precedes the others and additionally, medical or surgical interventions may result in serious side effects or complications. In 2005, the results of the Corticosteroid Randomization after Significant Head Injury (CRASH) trial raised concerns regarding the use of mega dose steroids in traumatic brain injury. This study was the largest randomized study that evaluated steroids in patients with traumatic brain injury and was stopped early due to the significantly increased risk of death in patients that received mega dose steroids at their 6-month follow-up when compared with the placebo group (25.7% vs 22.3%; Relative Risk 1.15 Confidence Interval 1.07 to 1.24; p=0.0001). Although the etiology of the increased risk of death was not determined, the findings of this study should be taken into consideration when managing cases of TON with concurrent traumatic brain injury. Very recently it has been shown the cytokine hormone erythropoietin (EPO) that had been long known and used as a valuable agent to promote hematopoiesis has been protective in experimental models of mechanical trauma, neuroinflammation, cerebral and retinal ischemia, and even in a human stroke trial, and most notably in optic nerve transection. A double blind placebo-controlled multicenter trial on EPO add-on treatment in chronic schizophrenic men was performed. Treatment over 12 weeks with high-dose weekly (40,000 IU intravenously) EPO led to significant improvement of cognitive performance compared to placebo controls. Different studies have been performed on the effect of EPO on neuropathy in different studies. The investigators recently published our results on treating patients with TON with EPO and found it safe and effective. Patients were compared with a historical control group of patients who received no treatment for TON. A better visual recovery was found. The aim of this study is to determine the effectiveness of EPO on TON in a Multi- center clinical trial using a semi-experimental design.

ELIGIBILITY:
Inclusion Criteria:

* Having indirect traumatic optic neuropathy, not more than 3 weeks between trauma and treatment, normal fundoscopy

Exclusion Criteria:

* Having other injuries that effect on visual function, direct optic neuropathy, glaucoma, diabetic retinopathy, uncontrolled hypertension, polycythemia, creatinin more than 3 mg/dl, sensitivity to EPO, hyperkalemia, women who use contraceptive pill, pregnant and breast feeding women, history of stroke and cardiovascular diseases, having malignancy

Ages: 5 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2015-02; Primary Completion 2016-04 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen B Kashkouli, MD, Study Chair — Iran University of Medical Sciences
Locations (3):
- Iran (3):
  - Shiraz University of Medical Sciences, Shiraz, Fars
  - Iran University of Medical Sciences, Tehran
  - Beheshti University of Medical Sciences, Tehran

RESULTS

PARTICIPANT FLOW:
Groups:
- Recombinant Human Erythropoietin (EPO): 20,000 unit per day of EPO, Intravenous infusion for three sequential days.
  Recombinant human erythropoietin (EPO): 4000 units per vial
- Methylprednisolone: 250 mg intravenous injection of Methylprednisolone for 3 days.
- Observation: No any treatment will be given
Period: Overall Study
Arm/Group | Recombinant Human Erythropoietin (EPO) | Methylprednisolone | Observation
Started | 85 | 16 | 16
Completed | 69 | 15 | 16
Not Completed | 16 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Methylprednisolone: 1 gram per day intravenous injection of Methylprednisolone for 3 days.
- Total: Total of all reporting groups
Arm/Group | Recombinant Human Erythropoietin (EPO) | Methylprednisolone | Observation | Total
Number analyzed (Participants) | 85 | 16 | 16 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 6 | 4 | 30
  Between 18 and 65 years | 64 | 10 | 12 | 86
  >=65 years | 1 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.4 (13.9) | 23.5 (9.4) | 29.0 (13.7) | 27.8 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 0 | 3 | 14
  Male | 74 | 16 | 13 | 103
Region of Enrollment [Number; unit: participants]
  Iran, Islamic Republic of | 85 | 16 | 16 | 117

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Change/Improvement Visual Acuity From the Beseline
Description: Best corrected visual acuity will measure at 1,2,3 days, 1 week, 2 weeks and 1 month and at least 3 months after treatment. Improvement is defined based on 1) mean logMAR[12], 2) 0.3 change in logMAR (improvement, deterioration, and no change) [12,16] , 3) mean improvement percentage which is calculated as: improvement%= (logMar ( of VA after treatment)-logMar ( of initial VA))/(logMar(20/13)˟-logMar ( of initial VA) 4) percentage of patients at different ordinal categorization of the BCVA as no light perception (NLP), light perception (LP)and hand motion (HM), count fingers (CF), and ≥ 20/200.
Time Frame: Change from baseline at least 3 months after treatment
Population: Seventeen patients with incomplete follow up and not following the treatment protocol were also excluded during the study. There were 100 patients (100 eyes) who completed the study protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Human Erythropoietin (EPO) | Methylprednisolone | Observation
Number analyzed (Participants) | 69 | 15 | 16
Participants | 28 | 3 | 5

2. Secondary Outcome: Number of Participants With Relative Afferent Papillary Defect (RAPD) Grade +4
Description: A positive RAPD means there are differences between the two eyes in the afferent pathway due to retinal or optic nerve disease. Graded from +1 to +4. The higher one is a better grade
Time Frame: Change from baseline at least 3 months after treatment
Population: Seventeen patients dropped out of the study due to incomplete follow-up (16 patients from EPO and one patient from Methylprednisolone group)
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Human Erythropoietin (EPO) | Methylprednisolone | Observation
Number analyzed (Participants) | 69 | 15 | 16
Participants | 26 | 7 | 8

ADVERSE EVENTS:
Arm/Group | Recombinant Human Erythropoietin (EPO) | Methylprednisolone | Observation
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 0/69 | 0/15 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes